CLINICAL TRIAL: NCT04408040
Title: Use of Convalescent Plasma Collected From Donors Recovered From COVID-19 Virus Disease for Transfusion, as an Empirical and Preemptive Treatment During Viral Pandemic Outbreak
Brief Title: Use of Convalescent Plasma for COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: New information regarding use of plasma in covid + patients
Sponsor: Northside Hospital, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSH 1281
Record Dates: First submitted 2020-05-15; First posted 2020-05-29 (Actual); Results first posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: COVID

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Critical Patients (Other)
  Interventions: Biological: Convalescent Plasma
- Severe Patients (Other)
  Interventions: Biological: Convalescent Plasma
- High Risk (Other)
  Interventions: Biological: Convalescent Plasma
- Health Care Providers (Other)
  Interventions: Biological: Convalescent Plasma

INTERVENTIONS:
Biological: Convalescent Plasma — 200-425mL convalescent plasma donated by patients previously positive for COVID-19

SUMMARY:
The plan is to transfuse COVID-19 infected patients with convalescent plasma and observe whether this will result in a significant improvement in clinical outcome in comparison to historical experience.

ELIGIBILITY:
Inclusion Criteria:

* Documented COVID-19 infection by nasal pharyngeal sampling
* COVID-19 disease falling into one of the following groups:
* Critical disease: respiratory failure requiring mechanical ventilation, pressor support, or multiple organ dysfunction/failure
* Severe disease: tachypnea >/=30 per min, O2 sats </=93% at rest, PaO2/FiO2 index </=300mmHg
* High Risk: upper respiratory symptoms but no radiographic evidence of disease, immunocompromised, insulin-dependent diabetes, poorly controlled HIV disease, moderate to severe asthma history, severe COPD, morbid obesity (BMI >/=40, age >/=65 years
* Health Care Providers: health care providers at risk to exposure to COVID-19 infection or those with mild to non-severe disease

Exclusion Criteria:

* History of IgA deficiency
* History of anaphylatic reaction to blood product transfusion including hypersensitivity to immunoglobulin therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kent Holland, MD, Principal Investigator — Northside Hospital
Locations (1):
- Northside Hospital, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period 7/14/2020-9/13/2021 Subjects were recruited from the hospital, outpatient clinic and from marketing efforts
Period: Overall Study
Arm/Group | Critical Patients | Severe Patients | High Risk | Health Care Providers
Started | 0 | 1 | 6 | 1
Completed | 0 | 1 | 6 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No critical patients were consented for this study
Groups:
- Total: Total of all reporting groups
Arm/Group | Critical Patients | Severe Patients | High Risk | Health Care Providers | Total
Number analyzed (Participants) | 0 | 1 | 6 | 1 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0 | 0 | 0
  Between 18 and 65 years |  | 1 | 5 | 1 | 7
  >=65 years |  | 0 | 1 | 0 | 1
Age, Continuous [Median (Full Range); unit: years] |  | 63 [63 to 63] | 37 [27 to 72] | 25 [25 to 25] | 37 [25 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 2 | 1 | 4
  Male |  | 0 | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0 | 0 | 0
  Asian |  | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0 | 0 | 0
  Black or African American |  | 0 | 3 | 0 | 3
  White |  | 1 | 3 | 1 | 5
  More than one race |  | 0 | 0 | 0 | 0
  Unknown or Not Reported |  | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 6 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Arms 1 & 2: Number of COVID-19 Infected Patients in Severe, High Risk & Health Care Provider Cohorts Who Survive the Infection
Description: Number of patients who survived the covid infection after treatment on study.
Time Frame: 30 days after initial treatment
Population: no critical patients were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Critical Patients | Severe Patients | High Risk | Health Care Providers
Number analyzed (Participants) | 0 | 1 | 6 | 1
Participants | 0 | 1 | 6 | 1

ADVERSE EVENTS:
Time Frame: 30 days
Description: 8 patients assessed
Arm/Group | Critical Patients | Severe Patients | High Risk | Health Care Providers
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1 | 0/6 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/6 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/6 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/40/NCT04408040/Prot_SAP_000.pdf